CLINICAL TRIAL: NCT07148128
Title: An Open-label, Multicenter, Phase 1/2a Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Antitumour Activity of WEF-001 in Participants With Advanced KRAS- Mutant Solid Tumours.
Brief Title: Phase 1/2a Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of WEF-001 as Monotherapy in Advanced KRAS-Mutant Solid Tumours.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Auricula Biosciences Inc. (Industry)
Collaborators: Simbec-Orion Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WEF-001-01; 2024-518644-21 (EudraCT Number)
Record Dates: First submitted 2025-06-25; First posted 2025-08-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Advanced or Metastatic KRAS-mutant Tumor in Pancreatic Adenocarcinoma; Advanced or Metastatic KRAS-mutant Tumor in Colorectal Cancer; Advanced or Metastatic KRAS-mutant Tumor in Non Small Cell Lung Cancer; Advanced Solid Tumors; Advanced or Metastatic KRAS-mutant Tumor
Keywords: Antineoplastic Agents; Advanced Solid Tumors; Pancreatic Cancer; Colorectal Cancer; KRAS Mutation-Related Tumors; Lung Cancer; Carcinoma, Non-Small Cell Lung Cancer; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Carcinoma; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose selection (Experimental): Phase 1: WEF-001 will be administered to participating patients at 1 selected dose out of 7 possible doses.
  Phase 2: WEF-001 will be administered to participating patients at 1 selected dose out of 2 possible doses.
  Interventions: Drug: WEF-001

INTERVENTIONS:
Drug: WEF-001 — Starting dose of 0.3 mg/m2 q4wks IV, dose escalation
  Other Names: MMAE-Drug Conjugate

SUMMARY:
This is a study designed to assess the safety, tolerability, pharmacokinetics and preliminary efficacy of WEF-001 as monotherapy in patients with Advanced KRAS-mutant solid tumours.

ELIGIBILITY:
Inclusion Criteria:

* Advanced KRAS-mutant solid tumor: pancreatic ductal adenocarcinoma, colorectal cancer, non small cell lung cancer, platinum-resistant serous ovarian cancer, cholangiocarcinoma or urothelial bladder cancer
* Progressive disease following at least one line of standard of care therapy
* Measurable disease as defined by RECIST v1.1
* ECOG ≤ 1

Exclusion Criteria:

* Active systemic infection requiring anti-infective therapy within 28 days prior to first dose of IMP
* Active cardiovascular disease
* Having a second active primary malignancy, requiring systemic administration of any cancer-related therapy
* Liver dysfunction
* Untreated brain metastasis and/or unstable neurological dysfunction
* Inflammatory bowel disease
* Active and untreated hyperthyroidism
* Lupus erythematosus within past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 110 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: To characterize the safety and tolerability profiles of WEF-001 administered as monotherapy. | Through study completion, an average of 1 year.
  Type, incidence and severity of TEAEs, SAEs and abnormal laboratory values per CTCAE v5.0.
  Frequency of dose interruptions, reductions, and discontinuations. Proportion of participants with DLTs at each dose level.
Phase 2: To evaluate the antitumour activity following WEF-001 administration as monotherapy. | Trough study completion, an average of 2 years.
  Objective Response Rate according to Response Evaluation Criteria in Solid Tumor (RECIST) v 1.1

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - NEXT Oncology Dallas, Dallas, Texas
  - Next Oncology, San Antonio, San Antonio, Texas
- Princess Margareth Cancer Center, Toronto, Ontario, Canada
- Oxford University Hospital, Headington, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No